CLINICAL TRIAL: NCT07132281
Title: A Language-Based Training Intervention to Enhance Cognitive Health in Community-Dwelling Older Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 202504009RIND
Record Dates: First submitted 2025-08-04; First posted 2025-08-20 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-07

CONDITIONS: Promoting Active Inference of Healthy Older Adults With Language Activity
Keywords: active inference; language; cognitive enhancement training; neuroscience; large language model
MeSH Terms: conditions — Language

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Active inference training (Experimental): Participants will undergo language activities and will be encouraged to actively infer based on the given language materials.
  Interventions: Behavioral: Language activities active inference
- Step-by-Step Guidance (Active Comparator): Participants will undergo language activities and will receive step-by-step guidance.
  Interventions: Behavioral: Language activities passive
- Board Games (Placebo Comparator): Participants will play boards games under a schedule matching the Experimental and Active Comparator arms.
  Interventions: Behavioral: Board Games

INTERVENTIONS:
Behavioral: Language activities active inference — Participants will join reading or writing activities and come up with their own inference about wording or plots.
  Arms: Active inference training
Behavioral: Language activities passive — Participants will join reading or writing activities and will be given step-by-step explanations about the wording and plots.
  Arms: Step-by-Step Guidance
Behavioral: Board Games — Participants will play board games with each other.
  Arms: Board Games

SUMMARY:
Taiwan is fast approaching a super-aged society, making it urgent to bolster cognitive health in otherwise healthy older adults. This integrated project tackles that need with a language-centered intervention grounded in predictive-coding and active-inference theory. Over 12 weeks, community-dwelling adults aged 65 + join small-group reading-and-writing workshops that train them to actively predict, monitor, and revise linguistic information. Ninety volunteers are randomly allocated to an active language-prediction group, a passive reading group, or a hobby board-game control. Before and after the course, researchers collect behavioural tests, EEG, fMRI, and AI-based speech-language analytics to quantify gains and transfer effects across cognition, emotion, and daily function.

DETAILED DESCRIPTION:
Taiwan will enter a super-aged society in 2025, with adults aged 65 and above expected to comprise 20 % of the population-a shift that makes preserving cognitive health an urgent public-health priority. To meet this challenge, our integrated project draws on predictive-coding and active-inference theory to couple language science with neuroscience, psychology, occupational therapy, and large-language-model analytics. Within this framework, the present sub-project tests a 12-week, small-group language-training curriculum that meets once a week for two hours. Sessions weave together reading aloud, listening, oral summarising, writing, and guided discussion, all structured to elicit continual prediction, self-monitoring, feedback, and creative revision during language use.

Approximately ninety community-dwelling adults aged 65 years or older are being recruited and randomly assigned, in equal blocks of thirty, to one of three arms: an active language-prediction group that emphasises hypothesis-testing during language production and comprehension; a passive reading group that provides leisure reading and sharing without explicit predictive feedback; and a board-game control group that engages cognition but not language prediction.

Before and after the intervention, each participant completes a comprehensive battery. Behaviourally, the investigators assess verbal fluency, language memory, and real-time sentence-prediction accuracy, while electrophysiology (N400, anterior-positivity ERPs, anterior P2, and P300) and functional MRI capture neural plasticity associated with sentence processing, visual reasoning, and cognitive flexibility. Executive functions, divergent and convergent thinking, attention, affect, social cognition, and instrumental activities of daily living provide secondary endpoints to gauge transfer beyond language. Throughout the 12 weeks, spoken narratives are recorded and analyzed for idea density and syntactic complexity with large-language-model tools, yielding fine-grained markers of change unavailable to traditional testing.

The investigators anticipate that targeted, prediction-based training will rejuvenate age-diminished language-prediction signals, drive adaptive reorganization of executive and language networks, and produce broader cognitive and functional gains than either passive reading or non-linguistic gaming. Embedded in community settings, this program also seeks to foster lasting reading habits, strengthen collective cognitive resilience, and offer an ecologically valid blueprint for scaling evidence-based cognitive-health interventions.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 20 and 30 (healthy young adults) or aged 65 and above (healthy older adults).
* Native Mandarin Chinese speakers who had no exposure to non-indigenous languages before the age of five.
* Have completed at least a junior high school level of education.
* Right-handed.
* Have normal or corrected-to-normal vision (e.g., through glasses or contact lenses).
* Able to fully participate in the entire assessment and intervention schedule (with no more than two missed intervention sessions).
* Achieve a score of 23 or higher on the Montreal Cognitive Assessment (MoCA).

Exclusion Criteria:

* Participation in another cognitive intervention program within the past two months.
* Cognitive intervention is not feasible due to dyslexia or physical illness. Meet the diagnostic criteria for Mild Cognitive Impairment (MCI) or dementia.
* Presence of severe depression, or cognitive changes caused by other psychiatric, neurological disorders, or substance abuse, with symptoms that are unstable or interfere with functioning.
* History of brain injury or neurological conditions (e.g., stroke, aneurysm).
* Contraindications for MRI scanning, such as metal implants, pacemakers, or pregnancy.
* Claustrophobia (an anxiety disorder characterized by panic symptoms or fear of panic attacks in enclosed spaces such as elevators, vehicles, tunnels, or airplane cabins).
* Unable to undergo cognitive assessments due to visual or hearing impairments.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-09-02 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes of neural functional activity during inferential processing | Week 0, Week 12
  Participants will undergo a Rule Inference fMRI task to infer underlying rules that map color configurations of circles in a triangular arrangement to a target color category within as few tries as possible under active or passive conditions. The goal for participants will be to infer the cue-category association rules using as few cues as possible. The primary outcome measure here is the degree of neural response estimate change in blood oxygen level dependent (BOLD) signal pre- and post-intervention.
Changes of overall accuracy during inferential processing | Week 0, Week 12
  Changes from pre- to post-intervention in participant overall accuracy in identifying latent rules in the Rule Inference fMRI task.
Changes of learning rate during inferential processing | Week 0, Week 12
  Changes from pre- to post-intervention in participant number of trials to criterion in the Rule Inference fMRI task.
Changes of strategic performance during inferential processing | Week 0, Week 12
  Changes from pre- to post-intervention in participant coefficients of expression of modeled response strategies in the Rule Inference fMRI task will be assessed.
Changes of functional electrical brain responses during reading | Week 0, Week 12
  Participants will undergo EEG language reading tasks in which participants were told to actively comprehend the sentence and to infer meanings for unknown pseudowords. The primary outcome measure here is the changes in N400 responses and anterior positive responses pre- and post-intervention.
Changes in the Montreal Cognitive Assessment (MoCA) score | Week 0, Week 12
  Pre- to post-intervention changes in participant MoCA score. Score range from 0 to 30 with higher scores indicating better cognitive ability.
Change in Wechsler Memory Scale III Logical Memory I & II | Week 0, Week 12
  Score range 0 - 75. Higher score indicates better verbal episodic memory.
Change in Wechsler Memory Scale III Face Memory | Week 0, Week 12
  Score range 0 - 48. Higher score indicates better visual face memory.
Change in Wechsler Memory Scale III Verbal Paired Memory | Week 0, Week 12
  Score range 0 - 32. Higher score indicates better verbal memory and learning.
Change in Wechsler Memory Scale III Family Pictures I & II | Week 0, Week 12
  Score range 0 - 64. Higher score indicates better visual memory and learning.
Change in Wechsler Memory Scale III Word Lists I & II | Week 0, Week 12
  Score range 0 - 36. Higher score indicates better verbal memory and learning. For II, recall score range is 0 to 8; recognition score range is 0 to 24.
Change in Wechsler Memory Scale III Visual Reproduction I & II | Week 0, Week 12
  Score range 0 - 104. Higher score indicates better visual memory. For II, recall score range is 0-104; recognition score range is 0-48.
Change in Wechsler Memory Scale III Spatial Span | Week 0, Week 12
  Score range 0 - 32. Higher score indicates better spatial memory.
Change in Wechsler Memory Scale III Digit Span | Week 0, Week 12
  Score range 0 - 32. Higher score indicates better auditory memory.
Change in Wechsler Adult Intelligence Scale III Vocabulary | Week 0, Week 12
  Score range 0 - 66. Higher score indicates better vocabulary.
Change in Wechsler Adult Intelligence Scale III Digit Symbol | Week 0, Week 12
  Score range 0 - 133. Higher score indicates better processing speed.
Change in Wechsler Adult Intelligence Scale III Block Design | Week 0, Week 12
  Score range 0 - 68. Higher score indicates better visual processing.
Change in Wechsler Adult Intelligence Scale III Arithmetic | Week 0, Week 12
  Score range 0 - 22. Higher score indicates better mathematical computation ability.
Change in Wechsler Adult Intelligence Scale III Matrix Reasoning | Week 0, Week 12
  Score range 0 - 26. Higher score indicates better reasoning.
Changes of overall accuracy for meaning inferences | Week 0, Week 12
  Changes from pre- to post-intervention in participants' overall accuracy in judging the semantic relation between newly learned pseudo-words and their semantic associates.
Changes of electrical brain responses during the task switching experiment | Week 0, Week 12
  Participants will undergo an EEG task-switching paradigm in which they are instructed to make an odd/even judgment or a size judgment on presented numbers.
Changes of overall accuracy during the task-switching paradigm | Week 0, Week 12
  Changes from pre- to post-intervention in participants' switch cost, assessed through overall accuracy.
Changes of Originality in Alternate Use Test (AUT) | Week 0, Week 12
  Developed by Guilford et al. (1967), this tool serves as a quantitative measure for assessing creativity and divergent thinking. In under three minutes, participants are given common multipurpose items and are asked to creatively think of uses for these items on paper, such as various uses for a brick. The scoring of Originality measures the uniqueness of the response in comparison to others. For instance, an answer that only 1% of participants come up with scores 2 points; an answer given by 5% scores 1 point.
Changes in Chinese Remote Association Task (CRAT) | Week 0, Week 12
  The Chinese Remote Association Task is used to measure individuals' abilities in convergent thinking. The original developer of the Remote Associates Test (RAT) was Mednick (1962). The Chinese version of the Remote Associates Test was developed by Huang et al. (2012). In this test, participants are provided with three Chinese words (e.g., Taiwan, land, barrier), and they are required to find a fourth Chinese word that forms a meaningful association with all three given words (e.g., strait). The study consists 30 questions and includes two versions of the test, A and B, which have a correlation of 0.610. The internal consistency coefficients for these versions are 0.808 and 0.801, respectively （Ren et al., 2004).
Changes of completion time in Color Trails Test (CTT) | Week 0, Week 12
  Performance is measured by recording the completion time.
Changes of number of trials administered in Wisconsin Card Sorting Test (WCST) | Week 0, Week 12
  Participants' performance is evaluated by measuring total trials required to complete the task (fewer trials indicate better performance).
Changes of overall fluency of language production | Week 0, Week 12
  Changes from pre- to post-intervention in participants' fluency in language production.
Changes of the number of errors in Color Trails Test (CTT) | Week 0, Week 12
  The Color Trails Test (CTT) is a neuropsychological assessment designed to measure sustained attention, alternating attention, and executive functioning (D'Elia et al., 1996). The test typically takes between 3 and 8 minutes to complete and consists of two parts. In Part 1, participants are instructed to connect numbered circles (1 through 25) in ascending order as quickly as possible. In Part 2, participants must again connect the numbered circles in order but are required to alternate between pink and yellow circles, adding a set-shifting and divided attention component. Performance is measured by the number of errors for each part. This study employed the Chinese adaptation of the CTT developed by Guo (2009), which includes normative data for Chinese adults aged 50 to 88 years. The test-retest reliability coefficients for Part 1 and Part 2 were reported as 0.618 and 0.833, respectively.
Changes of Fluency in Alternate Use Test (AUT) | Week 0, Week 12
  Developed by Guilford et al. (1967), this tool serves as a quantitative measure for assessing creativity and divergent thinking. In under three minutes, participants are given common multipurpose items and are asked to creatively think of uses for these items on paper, such as various uses for a brick. The scoring of Fluency measures the total number of responses.
Changes of Flexibility in Alternate Use Test (AUT) | Week 0, Week 12
  Developed by Guilford et al. (1967), this tool serves as a quantitative measure for assessing creativity and divergent thinking. In under three minutes, participants are given common multipurpose items and are asked to creatively think of uses for these items on paper, such as various uses for a brick. The scoring of flexibility is as follow: Responses are categorized based on their characteristics, and the number of categories is counted as the score.
Changes of overall reaction time during the task-switching paradigm | Week 0, Week 12
  Changes from pre- to post-intervention in participants' switch cost, assessed through overall reaction time.
Changes of percent correct in Wisconsin Card Sorting Test (WCST) | Week 0, Week 12
  The proportion of trials with correct responses is measured.
Changes of percent errors in Wisconsin Card Sorting Test (WCST) | Week 0, Week 12
  The proportion of trials with incorrect responses is measured.
Changes of number of categories completed in Wisconsin Card Sorting Test (WCST) | Week 0, Week 12
  The number of sorting categories completed is measured (i.e., 10 consecutive correct responses per rule).
Changes of trials to complete first category in Wisconsin Card Sorting Test (WCST) | Week 0, Week 12
  The number of trials required to achieve the first sorting criterion is measured.
Changes of percent perseverative responses in Wisconsin Card Sorting Test (WCST) | Week 0, Week 12
  The percent perseverative responses that continued to follow the previous rule, regardless of correctness, is measured.
Changes of percent perseverative errors in Wisconsin Card Sorting Test (WCST) | Week 0, Week 12
  The proportion of incorrect responses due to perseveration (i.e., failure to shift after rule change) is measured.
Changes of percent nonperseverative errors in Wisconsin Card Sorting Test (WCST) | Week 0, Week 12
  The proportion of incorrect responses not attributable to perseveration is measured.

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
Data that can be shared include anonymized neuropsychological assessment scores, cognitive behavioral performance scores, neurophysiological data that have been published.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Data will become available 1 year after primary results are published by the central research team. Data are anticipated to be available for sharing for an indefinite period after the above criteria is met.
Access Criteria: Data sharing will be done based direct requests and on case-by-case evaluation for appropriateness. Use of shared data will require agreement on appropriate citation of data sources at least or authorship inclusion or acknowledgement.